CLINICAL TRIAL: NCT02599662
Title: Phase I Study of Low Kilovoltage Intraoperative Radiation for Patients With Resectable Pancreatic Adenocarcinoma
Brief Title: Intraoperative Radiation Therapy for Resectable Pancreas Cancer
Acronym: IORT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Tarita Thomas, Assistant Professor of Radiation Oncology, Loyola University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 207194; 20719412115 (Other: Loyola University IRB)
Record Dates: First submitted 2015-11-05; First posted 2015-11-06 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Pancreas Cancer
Keywords: Cancer; Intraoperative Radiation Therapy - IORT
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1: 10 Gy Low-KV IORT (Other): 10 Gy Low Kilovoltage Intraoperative Radiation: intraoperative low-kV IORT will be delivered as a single dose of 10 Gy at 2 millimeter depth. Doses will be escalated in increments of 5 Gy until completion of 20 Gy dose level or the DLT is reached and MTD is realized.
  Interventions: Radiation: 10 Gy Low-KV IORT
- Group 2: 15 Gy Low-KV IORT (Other): 15 Gy Low Kilovoltage Intraoperative Radiation: intraoperative low-kV IORT will be delivered as a single dose of 15 Gy at 2 millimeter depth. Doses will be escalated in increments of 5 Gy until completion of 20 Gy dose level or the DLT is reached and MTD is realized.
  Interventions: Radiation: 15 Gy Low-KV IORT
- Group 3: 20 GY Low-KV IORT (Other): 20 GY Low Kilovoltage Intraoperative Radiation: intraoperative low-kV IORT will be delivered as a single dose of 20 Gy at 2 millimeter depth. Patients will be accrued to this group until the DLT is reached and MTD is realized.
  Interventions: Radiation: 20 GY Low-KV IORT

INTERVENTIONS:
Radiation: 10 Gy Low-KV IORT — : intraoperative low-kV IORT will be delivered as a single dose of 10 Gy at 2 millimeter depth. Doses will be escalated in increments of 5 Gy until completion of 20 Gy dose level or the DLT is reached and MTD is realized.
  Arms: Group 1: 10 Gy Low-KV IORT
Radiation: 15 Gy Low-KV IORT — intraoperative low-kV IORT will be delivered as a single dose of 15 Gy at 2 millimeter depth. Doses will be escalated in increments of 5 Gy until completion of 20 Gy dose level or the DLT is reached and MTD is realized.
  Arms: Group 2: 15 Gy Low-KV IORT
Radiation: 20 GY Low-KV IORT — intraoperative low-kV IORT will be delivered as a single dose of 20 Gy at 2 millimeter depth. Patients will be accrued to this group until the DLT is reached and MTD is realized.
  Arms: Group 3: 20 GY Low-KV IORT

SUMMARY:
Currently, for patients with pancreatic cancer the standard treatment is surgery followed by chemotherapy and/or radiation therapy. An investigational approach is to perform the surgery and treat the area of the tumor with intraoperative radiotherapy in one procedure. Intraoperative radiation delivers low energy x-rays to a targeted area during the time of tumor removal.

The purpose of this study is to learn about both the good and bad effects of adding intraoperative radiation therapy. Another goal is to determine and compare the quality of life before and after the procedure. We will also monitor the effect of the therapy on the cancer lesion and any complications that may result.

DETAILED DESCRIPTION:
The purpose of this study is to determine safety of low kilovoltage radiotherapy delivery of a focused dose of radiation to the areas at high risk for locoregional recurrence following pancreaticoduodenectomy. This surgery is currently the only potentially curative approach for patients with pancreatic cancer. Unfortunately, following surgery alone >50% of patients will have a local recurrence of disease [5]. Local control will become increasingly important as chemotherapy regimens continue to improve the distant metastases-free survival. Intraoperative radiation therapy allows direct access to the tumor bed and areas of concern while allowing displacement and shielding of normal tissue and organs at risk of radiation toxicity.

Study Objectives The primary objective is to determine the maximum tolerated dose (MTD) for low kilovoltage (kV) intraoperative radiotherapy (IORT)

The secondary objectives are:

To develop acute and chronic toxicity profiles for this treatment modality

To determine the feasibility of including low-kV IORT in the treatment of pancreatic cancer

To evaluate the following physics and delivery parameters: treatment prescription dose, depth of treatment, applicator type, and treatment time.

To measure patient's quality of life (QOL) before and after treatment, including change in pain level and fatigue level.

To describe the disease specific outcomes of local regional control, progression free-survival, distant metastasis free-survival, disease free-survival and overall survival associated with low-kV IORT following pancreaticoduodenectomy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed pancreatic adenocarcinoma.
* Age ≥ 18 years.
* Performance status ECOG 0-1.
* Patient must have resectable disease. In order to be resectable the following criteria must be met:
* Absence of distant metastases.
* Clear fat planes around the celiac axis, hepatic artery, and superior mesenteric artery .
* Absence of direct involvement of inferior vena cava or aorta.
* Stage I and stage II disease per AJCC 7th edition.
* Complete history and physical examination including weight and ECOG performance status within 31 days of entry.
* Laboratory data obtained ≤ 14 days prior to registration on study, with adequate bone marrow and organ function defined as follows:

Laboratory Test Result Leukocytes ≥3000/mm3 Absolute Neutrophil Count (ANC) ≥1500/mm3 Platelets ≥100,000/mm3 Total Bilirubin ≤1.4 mg/dL AST(SGOT),ALT(SPGT) ≤2.5 x institutional upper limit of normal Serum creatinine ≤1.4 mg/dL INR ≤1.5 BUN < 20 mg/dL Albumin ≥3.5 g/dL

* Negative serum pregnancy test for females of childbearing potential within 14 days of study registration. Should a female participant become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months.
* Abdominal CT scan with contrast prior to performance of surgery. If patient is allergic to contrast an abdominal MRI may substitute. Other imaging may be added or substituted as deemed appropriate by the treatment team (surgeon, radiation oncologist, medical oncologist).
* Ability to understand and the willingness to sign a written informed consent.
* Signed study specific informed consent.
* Patients with prior history of malignancy are permitted to register in the study as long as they are not actively taking cytotoxic or biologic medication for treatment of the prior malignancy. Patient must be disease-free from any malignancy for at least the previous 6 months and must have no history of brain metastases.
* Consultation, agreement, and documentation by a radiation oncologist that the patient is suitable to receive radiotherapy per this protocol.
* Consultation, agreement, and documentation by surgeon that the patient is a suitable surgical candidate.
* Consultation, agreement, and documentation by an anesthesiologist that patient is suitable to receive general anesthesia.

Exclusion Criteria:

* Defined treatment area which cannot be adequately covered by the radiation field as defined by the radiation oncology treatment team.
* Patients who have received neoadjuvant chemotherapy are ineligible.
* Patients with Stage III-Stage IV disease.
* Patients who have been on an immunosuppressive agent (excluding corticosteroids) within 4 weeks of the proposed operation.
* Patients receiving any other investigational agents.
* Current pregnancy or currently nursing.
* History of brain metastases.
* Severe, active comorbidity defined as follows
* Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months. [23]
* Myocardial infarction within 3 months of study registration [23].
* Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration.
* Chronic Obstructive Pulmonary Disease or other respiratory illness hospitalization or precluding study therapy at time of registration [23].
* Uncontrolled diabetes which in the opinion of any of the patient's physicians requires an immediate change in management. A patient may be considered eligible if the patient's physician managing the diabetes deems the appropriate changes in management have resulted in adequate control. [23].
* BMI >30.
* Patient with active diagnosis of a bleeding disorder. [23]
* Patients enrolled in another interventional clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-01; Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 52 weeks
  Maximum Tolerated Dose as defined by Radiation-related acute Grade 3-5 toxicity in greater than or equal to 2 patients out of 6 patients at any dose level

SECONDARY OUTCOMES:
QOL surveys | 52 weeks
  . The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQC30) 30 item questionnaire to evaluate cancer patients' physical, psychological, and social functioning. Patients are asked to rate symptoms on a YES or NO scale; a 4 point scale ranging from 1 (Not at all) to 4 (Very much); and a 7 point scale ranging 1 (Very poor) to 7 (Excellent)

CONTACTS AND LOCATIONS:
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

REFERENCES:
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2013. CA Cancer J Clin. 2013 Jan;63(1):11-30. doi: 10.3322/caac.21166. Epub 2013 Jan 17. PMID 23335087
- [Background] Kalser MH, Ellenberg SS. Pancreatic cancer. Adjuvant combined radiation and chemotherapy following curative resection. Arch Surg. 1985 Aug;120(8):899-903. doi: 10.1001/archsurg.1985.01390320023003. PMID 4015380
- [Background] Mohammed S, Van Buren G 2nd, Fisher WE. Pancreatic cancer: advances in treatment. World J Gastroenterol. 2014 Jul 28;20(28):9354-60. doi: 10.3748/wjg.v20.i28.9354. PMID 25071330
- [Background] Nagakawa T, Kayahara M, Ohta T, Ueno K, Konishi I, Miyazaki I. Patterns of neural and plexus invasion of human pancreatic cancer and experimental cancer. Int J Pancreatol. 1991 Oct;10(2):113-9. doi: 10.1007/BF02924114. PMID 1660909
- [Background] Gnerlich JL, Luka SR, Deshpande AD, Dubray BJ, Weir JS, Carpenter DH, Brunt EM, Strasberg SM, Hawkins WG, Linehan DC. Microscopic margins and patterns of treatment failure in resected pancreatic adenocarcinoma. Arch Surg. 2012 Aug;147(8):753-60. doi: 10.1001/archsurg.2012.1126. PMID 22911074
- [Background] Iqbal N, Lovegrove RE, Tilney HS, Abraham AT, Bhattacharya S, Tekkis PP, Kocher HM. A comparison of pancreaticoduodenectomy with extended pancreaticoduodenectomy: a meta-analysis of 1909 patients. Eur J Surg Oncol. 2009 Jan;35(1):79-86. doi: 10.1016/j.ejso.2008.01.002. Epub 2008 Mar 19. PMID 18356005
- [Background] Hiraoka T. Extended radical resection of cancer of the pancreas with intraoperative radiotherapy. Baillieres Clin Gastroenterol. 1990 Dec;4(4):985-93. doi: 10.1016/0950-3528(90)90031-b. No abstract available. PMID 2078795
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Wood WC, Shipley WU, Gunderson LL, Cohen AM, Nardi GL. Intraoperative irradiation for unresectable pancreatic carcinoma. Cancer. 1982 Mar 15;49(6):1272-5. doi: 10.1002/1097-0142(19820315)49:63.0.co;2-e. PMID 6800633
- [Background] Shipley WU, Wood WC, Tepper JE, Warshaw AL, Orlow EL, Kaufman SD, Battit GE, Nardi GL. Intraoperative electron beam irradiation for patients with unresectable pancreatic carcinoma. Ann Surg. 1984 Sep;200(3):289-96. doi: 10.1097/00000658-198409000-00006. PMID 6205632
- [Background] Kawai M, Yamaue H. Analysis of clinical trials evaluating complications after pancreaticoduodenectomy: a new era of pancreatic surgery. Surg Today. 2010 Nov;40(11):1011-7. doi: 10.1007/s00595-009-4245-9. Epub 2010 Nov 3. PMID 21046497
- [Background] Parikh P, Shiloach M, Cohen ME, Bilimoria KY, Ko CY, Hall BL, Pitt HA. Pancreatectomy risk calculator: an ACS-NSQIP resource. HPB (Oxford). 2010 Sep;12(7):488-97. doi: 10.1111/j.1477-2574.2010.00216.x. PMID 20815858
- [Background] Lermite E, Sommacale D, Piardi T, Arnaud JP, Sauvanet A, Dejong CH, Pessaux P. Complications after pancreatic resection: diagnosis, prevention and management. Clin Res Hepatol Gastroenterol. 2013 Jun;37(3):230-9. doi: 10.1016/j.clinre.2013.01.003. Epub 2013 Feb 14. PMID 23415988